CLINICAL TRIAL: NCT06317350
Title: A Prospective, Randomized, Parallel, Multi-center, Active Controlled, Single Blind (Assessor), Phase 3 Clinical Trial in Bowel Preparation for Colonoscopy
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of GNS-212-E in Bowel Preparation for Colonoscopy
Acronym: GNS-212-E
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gunkang Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GNS-212-E; 101772 (Other: MFDS)
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: colonoscopy; Bowel preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GNS-212-E1 (Experimental)
  Interventions: Drug: GNS-212-E1
- GNS-212-E2 (Experimental)
  Interventions: Drug: GNS-212-E2
- GNS-212-ER (Active Comparator)
  Interventions: Drug: GNS-212-ER

INTERVENTIONS:
Drug: GNS-212-E1 — Subjects who are randomized into this group will take GNS-212-E1 from the evening before colonoscopy to the morning of colonoscopy.
  Arms: GNS-212-E1
Drug: GNS-212-E2 — Subjects who are randomized into this group will take GNS-212-E2 from the evening before colonoscopy to the morning of colonoscopy.
  Arms: GNS-212-E2
Drug: GNS-212-ER — Subjects who are randomized into this group will take active control drug (PEG3350) from the evening before colonoscopy to the morning of colonoscopy.
  Arms: GNS-212-ER

SUMMARY:
This is a prospective, randomized, single-blind, parallel, active-controlled, and multi-center Phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women between 19 years and 79 age or older as of the date of consent in writing
2. 19 kg/㎡ ≤ BMI < 30 kg/㎡
3. a prospective colonoscopy patient
4. For women of childbearing potential, those who agree to use a medically acceptable contraceptive method* during the clinical trial period

   *hormonal contraceptive, implantation of intrauterine device or intrauterine system, Infertility procedures/surgery (e.g., bilateral ovarian ligation, vasectomy)
5. A person who voluntarily agrees to participate in this clinical trial and signs a written agreement Abbreviation
6. Women of childbearing potential must have a negative serum or urine pregnancy test before Investigational Product administration

Exclusion Criteria:

1. A person having constipation who is regularly administered laxatives or gastrointestinal motility promoters
2. A person with a history of significant gastrointestinal surgeries, including colonic resection, subtotal colectomy, abdominoperineal resection
3. A person diagnosed with acute coronary disease, arrhythmia, cardiomyopathy, cardiac valvular disease, aortic and peripheral vascular disease
4. Active infection or high fever above 38°C
5. Uncontrolled chronic medical illnesses or suspected symptoms that hinder participation such as major cardiac, renal, and metabolic (ex, Subjects with severe renal disease).
6. Clinically significant abnormal laboratory values of screening.(Creatinine, AST or ALT )
7. Active hepatitis B or hepatitis C with positive HBsAg and HCV Ab tests at screening
8. Positive for Human Immuno-deficiency Virus (HIV) at the time of screening
9. Severe nausea or vomiting
10. Severe abdominal distension or abdominal pain
11. A person prone to aspiration or reflux
12. A person who undergoes colonoscopy for the following therapeutic purpose (1) balloon dilatation of the stenosis area (2) non-toxic giant colon or decompression of the S-phase colitis (sigmoid volvulus) (3) Removal of foreign substances (4) Vascular dysplasia, ulcer, tumor and treatment of bleeding after polypectomy
13. A person who is hypersensitive to the ingredients of a clinical trial drug
14. Pregnant woman or a lactating woman
15. A person who has serious mental disabilities
16. A person who requires the administration of drugs prohibited from concomitant use
17. A person who is administered another investigational drug or has been provided with a clinical trial medical device within 6 months prior to participating in a clinical trial
18. The person whom the investigator determines to be unsuitable for this study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the successful % of bowel preparation before colonoscopy (colon cleanliness) using the HCS (Harefield Cleansing Scale) | on the day of scheduled colonoscopy
  HCS grading of A and B would be classified as successful while C and D would be classified as not successful

SECONDARY OUTCOMES:
Overall rate of bowel preparation | On the day of colonoscopy
  Percentage of test subjects for respective HCS grades
Overall patient satisfaction and compliance | before and on the day of colonoscopy
  Subject questionnaire evaluation total volume, taste etc.

CONTACTS AND LOCATIONS:
Overall Officials: Byeong Gwan Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea